CLINICAL TRIAL: NCT04483414
Title: The Role of 68Gallium PSMA-11 in Biochemical Recurrence in Prostate Cancer and in Known Metastatic Prostate Cancer and in the Evaluation of Treatment Response After Salvage Therapy
Brief Title: 68Ga PSMA-11 PET/CT in Recurrent Prostate Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was closed since no participants were enrolled.
Sponsor: Dana Mathews (Other)
Responsible Party: Sponsor-Investigator, Dana Mathews, Professor, University of Texas Southwestern Medical Center
Organization: University of Texas Southwestern Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STU-2020-0488
Record Dates: First submitted 2020-07-20; First posted 2020-07-23 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Prostate Cancer; Prostate Cancer Metastatic; Prostate Cancer Metastatic to Bone
Keywords: PET/CT; prostate cancer; Gallium-68; PSMA-11
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gallium 68 PSMA-11; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Intervention Model Description: Unblinded, single arm imaging study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Patients with suspected BCR or metastatic prostate cancer (Experimental): Patients with suspected BCR or metastatic prostate cancer
  Interventions: Drug: 68Ga PSMA-11 injection; Procedure: Positron Emission Tomography/Computed Tomography

INTERVENTIONS:
Drug: 68Ga PSMA-11 injection — Injection of 68Ga PSMA-11
Procedure: Positron Emission Tomography/Computed Tomography — PET/CT scan after 68Ga PSMA-11 injection
  Other Names: PET/CT

SUMMARY:
The goal of this research is to examine the ability of Gallium-68 (68Ga) Prostate-Specific Membrane Antigen-11 (PSMA-11) positron emission tomography/computed tomography (PET/CT) to detect sites of recurrent prostate cancer in patients with biochemical recurrence previously treated with radical prostatectomy (RP) or external beam radiation (EBRT) and to assess treatment response to subsequent salvage therapy.

DETAILED DESCRIPTION:
In developed countries, prostate cancer is the most common malignancy in men and the third leading cause of death in men. Following primary therapy for prostate cancer, a substantial number of patients will recur either locally in the pelvis or in extra pelvic locations. Approximately 20-30% of patients' status post RP will recur and up to 60% patients treated with EBRT will recur, as detected by rising serum levels of prostate specific antigen (PSA) after original therapy. This phenomenon is referred to as biochemical recurrence (BCR), as the elevated PSA usually occurs in advance of obvious clinical or radiologic evidence.

This study is designed to evaluate the performance of 68Ga PSMA-11 PET/CT in detecting the location (localized versus extra pelvic) of BCR and advanced metastatic prostate cancer compared to conventional imaging. In addition, we will evaluate its performance in assessing interim and post salvage therapy response compared to conventional imaging, including pelvic magnetic resonance imaging (MRI), computed tomography (CT), and bone scintigraphy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected BCR of prostate cancer following initial treatment with either prostatectomy or definitive EBRT of the prostate or patients with known metastatic prostate cancer who have failed systemic therapy.
* Patients being considered for salvage therapy.
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-3.
* Patients must be medically stable as judged by the patient's physician.
* Patients must be able to lie still for 20-40 minutes for the PET/CT scans.
* Ability to understand and the willingness to sign a written informed consent.
* Patients with BCR and no known lesions should not be on antiandrogen therapy at the time of scans. Patients with known metastases who are currently being treated with anti-androgen therapy may remain on this medication.

Exclusion Criteria:

* Patients who have or have had a biopsy proven concurrent other malignancy, excluding skin cancers.
* Patients may not weigh more than the maximum weight limit for the PET /CT scanner table (> 200 kg or 440 pounds).
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to 68Ga PSMA-11. Furosemide will not be administered to patients with known allergy.
* Patients must not be claustrophobic.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2021-03-19 (Actual); Primary Completion 2023-04-05 (Actual); Study Completion 2023-04-05 (Actual)

PRIMARY OUTCOMES:
Location of recurrence | Up to 3 years
  Localized vs extra-pelvic recurrence will be determined for each patient based on 68Ga PSMA-11 PET/CT and standard-of-care radiological imaging.
Residual prostate cancer | Up to 3 years
  For imaging during or after salvage therapy, existence of residual prostate cancer will be determined for each patient on 68Ga PSMA-11 PET/CT and standard-of-care radiological imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Orhan K Oz, MD, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No